CLINICAL TRIAL: NCT03892837
Title: Clinical Study on Autologous Platelet-rich Plasma (PRP) Treatment for Refractory Benign Airway Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Director of Department of Respiratory Medicine, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-03-06
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Benign Airway Stenosis
Keywords: Platelet-rich plasma; Refractory benign stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Procedure/Surgery: Conventional therapy of airway stenosis is including, but not limited to: laser, high frequency electric knife, argon plasma coagulation (APC), cryotherapy, balloon dilation and metal stent placement
  Interventions: Procedure: Conventional treatment for benign airway stenosis
- PRP group (Experimental): Procedure/Surgery: PRP PRP treatment following the conventional treatment Slow spray / inject autogenous PRP to cover the wound of stenosis. Procedure/Surgery: Conventional therapy of airway stenosis is including, but not limited to: laser, high frequency electric knife, argon plasma coagulation (APC), cryotherapy, balloon dilation and metal stent placement
  Interventions: Procedure: PRP; Procedure: Conventional treatment for benign airway stenosis

INTERVENTIONS:
Procedure: PRP — PRP treatment following the conventional treatment for benign airway stenosis which contain a concentrate of platelet-rich plasma protein derived from whole blood.
  Arms: PRP group
Procedure: Conventional treatment for benign airway stenosis — Including, but not limited to: laser, high frequency electric knife, argon plasma coagulation (APC), cryotherapy, balloon dilation and metal stent placement

SUMMARY:
Platelet-rich plasma(PRP), is a concentrate of platelet-rich plasma protein derived from whole blood. The main components of it are platelets, leukocytes and fibrin. Autologous PRP treatment can avoid the immune rejection caused by exogenous growth factor and the spread of disease. Evidence of the efficacy and safety of PRP has been proven in many studies. Benign central airway stenosis is characterized by airway compromise involving the larynx, trachea, or bronchi and will lead to devastating consequences. Unfortunately, the incidence of this disease is increasing steadily. As most important treatment for benign airway stenosis, respiratory intervention has become one of the most common treatments to fight the disease. However, the restenosis caused by tissue hyperplasia, wound repair and scar formation after treatment is still common, which remains the limitation of respiratory intervention. Long-term efficacy of repeated interventional treatment is unsatisfying, too. Several studies have discovered similar mechanism between stenosis of tracheal to hyperplastic scar of skin, both of which are relative with deep structure injury such as the intrinsic layer of airway mucosa. PRP has shown significant efficacy for hyperplastic scar of skin. Correspondingly, PRP will be applied as treatment of refractory benign airway stenosis to reduce restenosis by inhibit the formation of granulation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with aged between 18 to 75
2. Subjects diagnosed with refractory benign airway stenosis and meet the following conditions: a. Received two or more (including two) interventional treatments such as laser, high-frequency electrosurgical unit, argon plasma coagulation (APC), cryotherapy, balloon dilation, and metal stent placement. b. Restenosis within 1 month after more than 2 times interventional treatments suffering from repeated granulation hyperplasia of wound
3. Subjects tolerant to bronchoscope；
4. Subjects signed informed consent

Exclusion Criteria:

1. Subjects with airway disease:congenital benign central airway stenosis, recurrent polychondritis, etc;
2. Subjects with the following pulmonary diseases: asthma, active pulmonary tuberculosis, pulmonary embolism, pneumothorax, pulmonary hypertension, etc;
3. Subjects with malignant tumors or have a history of malignant tumors;
4. Subjects with uncontrolled systemic infection;
5. Subjects requiring anti-clotting drugs;
6. Subjects with myocardial infarction, unstable angina, liver cirrhosis, acute glomerulonephritis, etc;
7. Subjects with syphilis, HIV,HBV,HCV antibody positive;
8. Subjects with Coagulation disorders such as hemophilia, giant platelet syndrome, thromboasthenia, etc;
9. Subjects with severe renal damage, serum creatinine is more than 1.5 times the upper limit of the normal value;
10. Subjects with liver disease or liver damage: ALT,AST, total bilirubin > 2 times the upper limit of the normal value;
11. Subjects with a history of psychosis or suicide or epilepsy or other central nervous system diseases;
12. Subjects with severe arrhythmias(e.g. ventricular tachycardia, frequent supraventricular tachycardia, atrial fibrillation, atrial flutter, etc.) or degree II above abnormal conduction;
13. Subjects allergic to thrombin;
14. Subjects accepted by any other clinical study within the first three months of the study;
15. Subjects with poor compliance;
16. Any other conditions might increase the risk of the patient or interfere with the clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Cure rate for benign stenosis | within 6 months after administration
  Proportion of patients who is no need for endotracheal intervention and with stable clinical symptoms after PRP treatment

SECONDARY OUTCOMES:
Clinical remission time | 6 months after administration
  The interval time of the first intratracheal interventional therapy needed again after 6 times of PRP treatment
Times of unplanned treatment | within 6 months after administration
  The number of times a patient needs to be reviewed and treated by bronchoscopy for cough, expectoration and dyspnea
Incidence of complications associated with PRP treatment | within 6 months after administration
  Wound healing, sputum retention, etc. during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, MD, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No